Cover Page Study Title: Twitter and Cardiovascular Health NCT: NCT02806700

PI: Raina Merchant MD University of Pennsylvania

Re: Statistical analysis plan Last update 4.10.2018

Statistical Analysis Plan (Twitter and Cardiovascular Health:Twitter and Diabetes)

We will use summary statistics to compare demographics and survey responses (health status, ideal CV health status, self-practices) across groups. Summary statistics will be used to present data from the Perceived usefulness and Perceived ease of use measures for the intervention group.

For the primary and secondary outcome measures, we will use paired t-test for pre-post differences of scores. In addition, multivariable linear regression models will be used to model change in PAM score with adjustment for demographic and baseline health characteristics not evenly distributed by arm. In all models, a binary indicator for control/intervention group will be included. Baseline PAM score will also be adjusted for in the model. Covariates with missing data will be assessed for patterns of missingness and non-ignorability and will be multiply imputed if deemed necessary and reasonable.